CLINICAL TRIAL: NCT07067762
Title: Botulinum Toxin Injections in Salivary Glands of Brain-injured Children With Chronic Sialorrhea: a Retrospective Study.
Brief Title: Botulinum Toxin Injections Into the Salivary Glands of Cerebrospinal Children With Chronic Sialorrhea
Acronym: SIALOBOT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2025/961
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Drooling; Brain Injuries; Chronic Sialorrhea; Children, Only; Botulinum Toxin
MeSH Terms: conditions — Sialorrhea; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
French Health Authority describes sialorrhea (or drooling) as uncontrolled loss of saliva through the lips. Drooling is considered pathological after the age of three. It most often reflects an alteration in the control of orofacial muscular coordination. It is frequently observed in patients (adults and children) with neurological disorders. Among these neurological conditions, cerebral palsy is the most important cause of drooling in children. According to series, the incidence of drooling in children with cerebral palsy ranges from 10 to 58%, of whom 15% are considered to present with severe drooling.

Two types of drooling must be distinguished: anterior drooling (externalization of saliva through the lips) and posterior drooling (flow of saliva through the oropharynx that can reach the lungs by the trachea). Anterior drooling is responsible for skin erosions, fungal infections and dehydration, as well as low self-esteem and social rejection. Posterior sloughing, on the other hand, is not directly visible (unlike anterior sloughing).

Posterior bavage is not directly seen (unlike anterior bavage). However, should be noticed, as there is an increased risk of inhalation pneumonitis. Drooling is thus responsible for major social and emotional disturbances in affected children, as well as in parents/guardians/primary caregivers, justifying appropriate management. Many assessment tools are available to the clinician.

The subjective measures assess the social and emotional impact of daily life on patients and their families. For example, the Drooling Impact Scale (D.I.S.) was created by the salivary control department at Melbourne Hospital, Australia to add a subjective dimension to scales that do not assess the daily impact of drooling. There is no currently consensus method for assessing drooling importance or severity

Lot of treatment cas be proposed to patients with chornic sialorrheaalorrhea: non-drug treatments, medication (systemic or focal) and surgical treatments. Non-drug treatments consist of targeted rehabilitation by speech therapists and dental care. There is a wide range of rehabilitation techniques. However, this rehabilitation can only be effective in patients with the appropriate cognitive functions to enable them to understand and continue the exercises. Currently, there is little evidence of the effectiveness of these techniques in the scientific literature. Medication are used for their anticholinergic effect. However, due to their non-selective effect and systemic effects, medication are frequently associated with severe side-effects. These are sometimes more serious than sialorrhea, which limits the use of these molecules.

Botulinum toxin, injected specifically in the main salivary glands, has been used to treat drooling since 1997, thanks to its focal anticholinergic effect. Its efficacy has been demonstrated by randomized clinical trials: botulinum toxin has been shown to significantly reduce the frequency and severity of drooling. However, few studies have looked specifically at the efficacy of botulinum toxin in children in terms of functional and social repercussions using a subjective measurement scale.

The aim of the SIALOBOT study was to demonstrate the efficacy of botulinum toxin in the salivary glands of children with chronic sialorrhea, according to a subjective measure of daily functional impact

ELIGIBILITY:
Inclusion Criteria:

* Brain injured children aged 3 to 15, treated in the PRM department of Besançon University Hospital between 2021 and 2025, with chronic invalidating Sialorrhea for more than three months at the time of treatment, treated with botulinum toxin injections in the salivary glands.
* Minimal weight of 12 kg,
* Stopped drooling treatments three months before injections,
* Subject (holders of parental authority) does not refuse the use of personal data
* Registration with French social security plan.

Exclusion Criteria:

* Previous treatment with botulinum toxin in the salivary glands,
* Treatment with botulinum toxin for another indication in the previous three months,
* Contraindication to botulinum toxin injections.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: brain-injured children from 3 to 15 years of age with chronic sialorrhea.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2025-05-19 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of botulinum toxin in the treatment of drooling | Five weeks
  Use of the drooling impact scale to measure the efficacy of botulinum toxin on the frequency, severity and daily impact of drooling in brain injured children with chronic sialorrhea Each question is answered on a visual analogue scale (1-10) giving a score/100. 100 is the worst score (drooling had worsened).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Jean-Minjoz, Besançon, France